CLINICAL TRIAL: NCT03110913
Title: Study Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Methionine From Canadian Lentils, in Healthy Young Adult Men
Brief Title: Metabolic Availability of Metionine From Lentils in Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Project Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000056244
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Healthy
Keywords: Healthy; Men; Adults; Methionine
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Eating

STUDY DESIGN:
Intervention Model Description: Each subject will randomly receive 4 levels of methionine provided as free amino acids, lentils, or lentils combined with rice for a total of 10 studies x 3 days per study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methionine bioavailability in lentils (Experimental): Participants will be seen initially for pre-study assessment (3 hour). They will then be studied for up to 10 times. levels of phenylalanine intake (7 Study periods).
  You could be expected to participate in up to 10 different sets of experiments which will take 11 weeks to 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein free-cookies and/or a lentil stew with or without rice, which will be provided by the investigators
  Interventions: Other: dietary intakes

INTERVENTIONS:
Other: dietary intakes — Four levels of methionine intakes will be provided by the reference protein drinks, 3 levels of methionine from lentils and 3 levels from lentils with rice.

SUMMARY:
The research study is being done so we can determine the quality of the protein present in Canadian lentils. Amino acids are the building blocks of protein and protein quality is determined by the amount of amino acids present and by their bioavailability (their absorption and use by the body). Some amino acids are essential which means they must be obtained from the diet. If any one of the essential amino acids is missing in the diet, the body cannot make proteins that are used to repair tissue build bone, teeth, etc… Lentils as a food source contain low amounts of the essential amino acid methionine which makes its protein incomplete. The amino acids in lentils are also affected by cooking. Our objective is to determine the amount of methionine in lentils that the body can use. We will test lentils by studying them after cooking them in a stew, on their own and by combining the lentil stew with rice in a mixed meal to make a more complete protein.

This research is being done in order to bridge the gap between knowledge of protein requirement and the amount of food needed to meet that requirement. Results from this study will be important for recommendations guiding food choices of lentils as a major protein source in the diet.

Previously the quality of dietary protein for human consumption was studied in animals. This study is being done in humans because studies in animals are not directly applicable to humans. Excessive animal protein consumption is also linked to cardiovascular disease. Plant protein sources like lentils are important alternatives shown to "enhance ecosystem resilience, and improve human health.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will receive 3 different amounts of lentils which will contain different amounts of the essential amino acid methionine as well as 3 different amount of lentils complemented with rice. The lentils will be cooked in a stew served on its own or served with the rice. The quality of the protein in the lentils will be compared to the quality of a reference protein (egg protein) by giving you 4 reference diets containing amino acids make up like the amino acids in egg protein. The amount of lentils you receive will be provided in a random order.

Breath samples will be collected after the 4th meal in 15 min intervals for 1 hour. Breath collection will resume again two and a half hours after the 5th meal every 15 minutes until 30 minutes after the last meal. A total of 52 breath samples will be collected during each of the 3rd study day.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18 - 49 yrs, Healthy with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes, Stable Body Weight (no more than 5 lb weight loss or gain in the past 3 months) Not on any medications that could affect protein or amino acid metabolism e.g. steroids

Exclusion Criteria:

* Unwillingness to participate or unable to tolerate the diet Recent history of weight loss within the last 3 months or on a weight reducing diet Inability to tolerate study diets (ex. Allergy to ingredients).

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Metabolic availability of methionine in Canadian lentils | 2 years
  Apply the IAAO method to determine the MA of methionine in Canadian grown lentils prepared by moist cooking method.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rafii M, Pencharz PB, Boileau K, Ball RO, Tomlinson C, Elango R, Courtney-Martin G. Metabolic Availability of Methionine Assessed Using Indicator Amino Acid Oxidation Method, Is Greater when Cooked Lentils and Steamed Rice Are Combined in the Diet of Healthy Young Men. J Nutr. 2022 Jun 9;152(6):1467-1475. doi: 10.1093/jn/nxac049. PMID 35218191